CLINICAL TRIAL: NCT03877211
Title: Impact of Channel Interaction on Cochlear Implant Performances in Noise : Influence of the Number of Maxima.
Brief Title: Channel Interaction in Cochlear Implant and Speech Understanding in Noise
Acronym: 2IPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0434
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2022-03

CONDITIONS: Cochlear Implants
Keywords: speech audiometry; psychophysical tuning curve; electrophysiology; auditory brainstem response
MeSH Terms: interventions — Noise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cochlear implant users (Experimental): Adult cochlear implanted patients wearing an Oticon Medical/Neurelec device will have speech audiometry test in noise, psychophysical tuning curves in forward masking and Electrically-evoked Auditory Brainstem Response (EABR) measurement
  Interventions: Other: speech audiometry in noise; Other: Psychophysical tuning curves in forward masking; Other: Electrically-evoked Auditory Brainstem Response (EABR)
- Normal-hearing subjects (Active Comparator): Normal-hearing subjects will have speech audiometry test in noise, psychophysical tuning curves in forward masking, auditory canal examination and tonal audiometry
  Interventions: Other: speech audiometry in noise; Other: Psychophysical tuning curves in forward masking; Other: Tonal audiometry; Other: Auditory canal examination

INTERVENTIONS:
Other: speech audiometry in noise — Subjects will be asked to repeat lists of words played by speakers in a noisy environment generated by the same speakers. A percentage of correct recognition is calculated for each list.
Other: Psychophysical tuning curves in forward masking — Sounds of variable center frequency are used as maskers, and a tone with a fixed frequency at a fixed level is the target. What is tested here is the level of masker that just masks the target.
Other: Electrically-evoked Auditory Brainstem Response (EABR) — Channel interaction assessment using eABRs (auditory nerve responses). The method consists of two measurements: 1) eABR measurements with stimulation by a single electrode of the cochlear implant at 70% of the dynamic range (four different electrodes are tested); 2) Measurement of a single eABR with stimulation from all four electrodes at 70% of the dynamic range. A comparison of the eABRs obtained by these two measurements, indicates the electrical and neural interactions between the electrodes.
  Arms: Cochlear implant users
Other: Tonal audiometry — Tonal audiometry will be performed with headphones
  Arms: Normal-hearing subjects
Other: Auditory canal examination — Otoscopic examination of external auditory canal and eardrum
  Arms: Normal-hearing subjects

SUMMARY:
The goal of this study is to take into account channel interaction in the cochlear implant (CI) fitting process. Designing a fast and accurate method of measurement would help to customize the fitting procedures to patients' specificities in order to maximize speech understanding in every day conditions especially in noise.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in French
* Able to understand written instructions
* Under French public medical insurance

  * Normal-hearing subjects only:

    * Adult between 18 and 50 years old
    * Without a remarkable otological medical history, for example: chronic otitis, trans-tympanic tubes and / or all ear surgeries;
    * Clear auditory canal and normal eardrum;
    * Average audiometric loss under 20 decibels Hearing Level (dB HL)
  * Cochlear implant users only:

    * Adult between 18 and 60 yo
    * Normal middle ear
    * Used the cochlear implant for more than a year
    * Wearing a device from the company Neurelec/Oticon Medical

Exclusion Criteria:

* Behavioral and/or neurological disorders
* Proven psychological disorder
* Use of psychotropic medication
* People who experience migraine attacks on a regular basis
* Use of ototoxic medication
* Exposed to loud noises within the last 72 hours
* Included in another clinical trial that uses medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-24 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Percentage of syllable correctly recognized during speech audiometry test | At inclusion
  Subjects will be asked to repeat lists of words played by speakers in a noisy environment generated by the same speakers. A percentage of correct recognition is calculated for each list.

SECONDARY OUTCOMES:
Sound masking threshold | At inclusion
  Measurement of channel interaction by establishing psychophysical tuning curves in forward masking. Sounds of variable center frequency are used as a masker, and a tone with a fixed frequency at a fixed level is the target. What is tested here is the level of masker that just masks the target.
Electrically-evoked Auditory Brainstem Response (eABR) | Up to 12 months after inclusion
  Channel interaction assessment using eABRs (auditory nerve responses). The method consists of two measurements: 1) eABR measurements with stimulation by a single electrode of the cochlear implant at 70% of the dynamic range (four different electrodes are tested); 2) Measurement of a single eABR with stimulation from all four electrodes at 70% of the dynamic range. A comparison of the eABRs obtained by these two measurements, indicates the electrical and neural interactions between the electrodes.

CONTACTS AND LOCATIONS:
Overall Officials: Eric TRUY, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- ENT and Cervico-Facial Surgery Department, Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cucis PA, Berger-Vachon C, Thai-Van H, Hermann R, Gallego S, Truy E. Word Recognition and Frequency Selectivity in Cochlear Implant Simulation: Effect of Channel Interaction. J Clin Med. 2021 Feb 10;10(4):679. doi: 10.3390/jcm10040679. PMID 33578696